CLINICAL TRIAL: NCT01811784
Title: A Community Intervention Trial Utilizing Behavior Change to Reduce the Risk of Nipah Spillover Through Date Palm Sap in Bangladesh
Brief Title: Community Intervention to Prevent Nipah Spillover
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: FHI 360 (Other); IEDCR, DGHS, Bangladesh (Unknown); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-12053
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-02

CONDITIONS: Human NiV Infection
Keywords: Nipah virus infection; date palm sap; community intervention; capacity building; disease prevention; Bangladesh; Healthy Community people; Sap harvesters; Date palm three owners; Date palm sap consumers
MeSH Terms: conditions — Henipavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Use skirt on raw sap consumption (Experimental): Phase one: Test the effectiveness of a single message of "do not drink raw sap".
  Interventions: Behavioral: Ask people not to drink raw sap; Other: No Intervention
- Ask people not to drink sap (Experimental): Test the effectiveness of a risk reduction approach, encouraging people to avoid drinking sap, if they do, they should only drink sap from skirt protected trees.
  Interventions: Behavioral: Ask people not to drink sap or drink sap from skirt protected trees; Other: No Intervention
- Phase 1: Routine raw sap consumption among household members. (No Intervention): Test the effectiveness of a single message of "do not drink raw sap"
- Phase 2: (No Intervention): Raw sap consumption from skirt protected trees

INTERVENTIONS:
Behavioral: Ask people not to drink raw sap
  Arms: Use skirt on raw sap consumption
Behavioral: Ask people not to drink sap or drink sap from skirt protected trees — Behavioural
  Arms: Ask people not to drink sap
Other: No Intervention
  Arms: Use skirt on raw sap consumption
Other: No Intervention
  Arms: Ask people not to drink sap

SUMMARY:
Several human Nipah virus (NiV) outbreaks have occurred in Bangladesh since 2001with 71% case fatality. Outbreak investigations have repeatedly identified drinking fresh date palm sap as a risk factor for NiV transmission. Bats are the reservoir of NiV and infected bats can shed virus through both saliva and urine and can contaminate the raw sap. The virus can transmit to humans through ingestion of contaminated sap. To interrupt bats access to the sap, sap harvesters (gachhis) occasionally use skirts make by local materials. These skirts have been found to be effective to interrupt bats' access to the sap. As an indirect effect of the community level skirt promotion, some people stopped drinking raw sap. When trees have skirts, bats cannot access the sap and when people do not drink sap, they are at much lower risk of contracting Nipah virus. The purpose of this study is to design, implement and evaluate behavior change interventions to prevent human consumption of NiV contaminated sap through reducing raw sap consumption from unprotected trees in a district of the NiV affected regions in Bangladesh.

DETAILED DESCRIPTION:
Purpose:

Objectives: To evaluate the effectiveness of a behavior change communication (BCC) intervention in changing raw sap consumption behavior to prevent human consumption of NiV contaminated sap from unprotected trees in the districts of Rajbari (Phase one) and Natore (Phase two), in NiV-affected regions in Bangladesh.

Methods: The research study will be conducted in two phases.

Phase one:

We will conduct a BCC program to test the effectiveness of a single message of "do not drink raw sap". We will conduct a baseline survey as pre-intervention assessment in two intervention upazillas in Rajbari District and two control upazillas in Kushtia District. The intervention will consist of community meetings in each of the intervention area villages as well as an awareness campaign through closed circuit television in selected village tea stalls. We will conduct endline survey to as a post intervention assessment in the same upazillas in Rajbari and Kushtia Districts.

Main outcome measures/variables: Proportion of people who continue drinking raw date palm sap.

Phase two If a substantial proportion of the population continues to consume raw date palm sap even after implementation of the "avoid drinking sap" intervention, and the Government of Bangladesh agrees, we will conduct a BCC program to test the effectiveness of a risk reduction approach, encouraging people to avoid drinking sap, but telling them that if they do, to reduce risk they should only drink sap that comes from trees protected by banas. In addition to community meetings to convey this message to the general public, we will meet with gachhis and tree owners to encourage them to use banas. We will conduct a baseline survey as pre-intervention assessment in both intervention and control areas in Natore and Gopalganj Districts respectively. The intervention will consist of meetings with gachhis, tree owners and the community in each of the intervention area villages as well as an awareness campaign through closed circuit television in village tea stalls. We will conduct endline survey to as a post intervention assessment in both intervention (Natore District) and control areas (Gopalganj District).

Main outcome measures/variables: Proportion of people who stop drinking sap or who drink sap from skirt protected trees.

ELIGIBILITY:
Inclusion Criteria:

For baseline and endline:

* Women: the wife of the main male income earner in the household.
* Men: the main income earner.
* Sap harvesters.

Exclusion Criteria:

* If the desired respondent is not in the household the team will make an appointment to return to the household. If the desired respondent will not be available within 24 hours, the household will be skipped.
* Household visitors.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7782 (Estimated)
Dates: Start 2012-11-10 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Phase one: Proportion of people who continue drinking raw date palm sap. | 16 months
Phase two: Proportion of people who stop drinking sap or who drink sap from skirt protected trees. | 10 months

SECONDARY OUTCOMES:
Reduce human exposure to Nipah virus thought bat contaminated sap and increase the awareness level on prevention of Nipah virus by refraining from sap consumption. | 16 months

CONTACTS AND LOCATIONS:
Locations (4):
- Bangladesh (4):
  - Two sub-districts in Gopalganj, Gopālganj
  - Mirpur and Bheramara, Kushtia
  - two sub-districts in Natore, Natore
  - Pangsha and Kalukhali sub-districts, Rājbāri